CLINICAL TRIAL: NCT04900181
Title: Analysis of the Cost-Effectiveness of Same-day Discharge Surgery for Primary Total Hip Arthroplasty: A Pragmatic Randomized Controlled Study
Brief Title: Analysis of the Cost-Effectiveness of Same-day Discharge Surgery for Primary Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271816
Record Dates: First submitted 2021-03-29; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Hip Arthropathy
Keywords: same-day discharge surgery; total hip arthropathy; cost effectiveness

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the same-day discharge surgery (Experimental): Patients in the the same-day discharge surgery group were admitted to hospital, operated and discharged within 24 hour
  Interventions: Procedure: the same-day discharge surgery
- inpatient surgery (No Intervention): Patients in inpatient surgery follow routine procedures and do not need to be discharged on the same day.

INTERVENTIONS:
Procedure: the same-day discharge surgery — the same-day discharge surgery is the procedure in which the patient is admitted, operated and discharged within 24 hours.
  Arms: the same-day discharge surgery

SUMMARY:
Total hip arthroplasty (THA) causes a great medical burden globally, and the same-day discharge (SDD) method has previously been considered to be cost saving. However, a standard cost-effectiveness analysis (CEA) in a randomized controlled trial (RCT) is needed to evaluated the benefits of SDD when performing THA from the perspective of both economic and clinical outcomes. So the objective is to evaluate the cost-effectiveness of SDD for hip replacement.

This was a single center, pragmatic RCT with a 6-month follow up. Eighty-four participants who met the inclusion criteria were randomized to either the SDD group or the inpatient group (42 per group). Outcomes were assessed by an independent orthopedist who was not in the surgical team, using the Oxford Hip Score (OHS), EuroQol 5D (EQ-5D) and 36-Item Short-From Health Survey (SF-36) scores at the baseline and the 6-month follow up. All interviews were conducted face to face. All the cost information was collected both from payment receipts and insurance reimbursement records.

DETAILED DESCRIPTION:
This was a prospective RCT. Patients qualified for inclusion in the study if they met the following criteria: undergoing unilateral primary THA; having the ability to understand the relevant treatment process; aged between 18 and 75 years; a body mass index (BMI) ≤ 40 kg/m2; hemoglobin ≥ 12g/dL; American Society of Anesthesiologists (ASA) physical status classification of I or II; and no ongoing infection or blood coagulation disorders. Those with a history of coronary artery disease, chronic obstructive pulmonary disease, arrhythmias, or untreated obstructive sleep apnea were excluded. Eligible individuals who gave informed consent were randomly assigned (1:1) to an inpatient THA group or an SDD THA group. SDD-THA was defined as admission, surgery, and discharge within 24 hours, whereas the inpatients stayed in hospital for more than one day. Randomization occurred at the individual level and was performed by an independent statistician, utilizing an automatic computer-generated table of random numbers. Preoperatively, patients undergoing SDD-THA and their families received information in the form of teaching booklets and a teaching class conducted by a bedside clinician, which included the protocol, matters needing attention, exercise training, and home-based rehabilitation. All operations were performed by the same surgical team through a posterolateral approach. Standardized general anesthesia was administered by low-dose bupivacaine, to allow early postoperative patient mobilization. Celebrex 400 mg PO was used as routine analgesia before surgery. Cefazolin (1.0 g) and Tranexamic Acid (0.4 g) were administered 30 min prior to skin incision. A uniform perioperative multimodal pain management protocol was established by cocktail periarticular injection before wound closure, which consisted of Flurbiprofen axetil (50 mg) and Ropivacaine (200 mg). Patients in both groups accepted the same postoperative protocols. To avoid venous thromboembolism (VTE), all participants were encouraged to perform ankle pumping and quadriceps-setting exercises immediately. Additionally, patients were encouraged to get out of bed and ambulate progressively with assistance under the guidance of the bedside clinician.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral primary THA
* having the ability to understand the relevant treatment process
* aged between 18 and 75 years
* a body mass index (BMI) ≤ 40 kg/m2
* hemoglobin ≥ 12g/dL
* American Society of Anesthesiologists (ASA) physical status classification of I or II
* no ongoing infection or blood coagulation disorders

Exclusion Criteria:

* with a history of coronary artery disease
* chronic obstructive pulmonary disease
* arrhythmias
* untreated obstructive sleep apnea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
the Oxford Hip Score | six months
  the Oxford Hip Score consists of 12 questions reflecting the different aspects of hip function. Each question was scored from 0 to 4, with 4 representing the best outcome or least symptoms

SECONDARY OUTCOMES:
the quality-adjusted life years | six months
  the quality-adjusted life years was calculated as the outcome in cost utility analysis, as proposed by the CHEERS and CEA guidelines. The values of QALYs were estimated by EQ-5D . The EQ-5D was administered at baseline and at the 6-month follow-up. The EQ-5D is divided into five aspects (mobility, self-care, usual activities, discomfort, depression) to evaluate patients' health state, and each consists of three levels. The score for the EQ-5D ranges from -0.59 to 1.00, with a higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Tian, doctor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurtz SM, Ong KL, Lau E, Bozic KJ. Impact of the economic downturn on total joint replacement demand in the United States: updated projections to 2021. J Bone Joint Surg Am. 2014 Apr 16;96(8):624-30. doi: 10.2106/JBJS.M.00285. PMID 24740658
- [Result] Molloy IB, Martin BI, Moschetti WE, Jevsevar DS. Effects of the Length of Stay on the Cost of Total Knee and Total Hip Arthroplasty from 2002 to 2013. J Bone Joint Surg Am. 2017 Mar 1;99(5):402-407. doi: 10.2106/JBJS.16.00019. PMID 28244911
- [Result] Navathe AS, Troxel AB, Liao JM, Nan N, Zhu J, Zhong W, Emanuel EJ. Cost of Joint Replacement Using Bundled Payment Models. JAMA Intern Med. 2017 Feb 1;177(2):214-222. doi: 10.1001/jamainternmed.2016.8263. PMID 28055062
- [Result] Doran JP, Zabinski SJ. Bundled payment initiatives for Medicare and non-Medicare total joint arthroplasty patients at a community hospital: bundles in the real world. J Arthroplasty. 2015 Mar;30(3):353-5. doi: 10.1016/j.arth.2015.01.035. Epub 2015 Jan 23. PMID 25680450
- [Result] Zeng JQ. The pilot results of 47 148 cases of BJ-DRGs-based payment in China. Int J Health Plann Manage. 2019 Oct;34(4):1386-1398. doi: 10.1002/hpm.2818. Epub 2019 Jul 8. PMID 31286577
- See also: The link of citation — http://pubmed.ncbi.nlm.nih.gov/